CLINICAL TRIAL: NCT01088789
Title: A Safety and Feasibility Trial of Boost Vaccinations of a Lethally Irradiated, Allogeneic Pancreatic Tumor Cell Vaccine Transfected With the GM-CSF Gene Given Alone or in Combination With Either a Single Intravenous Dose or Daily Metronomic Oral Doses of Cyclophosphamide for the Treatment of Surgically Resected Pancreatic Adenocarcinoma
Brief Title: Boost GVAX Pancreas Vaccine With or Without CY in Patients With Pancreas Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Skip Viragh Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J09100; NA_00031401 (Other: JHM IRB)
Record Dates: First submitted 2010-03-01; First posted 2010-03-17 (Estimated); Results first posted 2025-07-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
Keywords: Adenocarcinoma; Cyclophosphamide; Immunotherapy; Adjuvant; Pancreatic tumor vaccine; GM-CSF; GVAX; Cancer vaccine
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 (J0810 Arm A) (Experimental): Patients coming from J0810 (NCT00727441). Patients receive GVAX.
  Interventions: Biological: GVAX Pancreas Vaccine
- Cohort 1 (J0810 Arm B) (Experimental): Patients coming from J0810 (NCT00727441). Patients receive IV CY and GVAX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Cohort 1 (J0810 Arm C) (Experimental): Patients coming from J0810 (NCT00727441). Patients receive oral CY and GVAX.
  Interventions: Drug: Cyclophosphamide Pill; Biological: GVAX Pancreas Vaccine
- Cohort 2 (Vaccine Naive) (Experimental): Patients receive IV CY and GVAX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Cohort 3 (J1568) (Experimental): Patients coming from J1568 (NCT02451982). Patients receive IV CY and GVAX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Cohort 4 (J15237) (Experimental): Patients coming from J15237 (NCT02648282). Patients receive IV CY and GVAX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine
- Cohort 5 (J1766) (Experimental): Patients coming from J1766 (NCT03153410). Patients receive IV CY and GVAX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine

INTERVENTIONS:
Drug: Cyclophosphamide — Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  Other Names: CY
  Arms: Cohort 1 (J0810 Arm B); Cohort 2 (Vaccine Naive); Cohort 3 (J1568); Cohort 4 (J15237); Cohort 5 (J1766)
Drug: Cyclophosphamide Pill — Cohort 1 patients (J0810 Arm C) will receive 50mg oral CY once a day starting 28 days prior to GVAX and for 28 days post-GVAX (every 6 months).
  Other Names: CY
  Arms: Cohort 1 (J0810 Arm C)
Biological: GVAX Pancreas Vaccine — Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
  Other Names: Panc 10.05 pcDNA-1/GM-Neo, Panc 6.03 pcDNA-1/GM-Neo

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of long term boost vaccination of a lethally irradiated, allogenic pancreatic tumor cell vaccine transfected with the granulocyte macrophage colony-stimulating factor (GM-CSF) gene (GVAX Pancreas Vaccine) alone or given in combination with either a single intravenous dose or daily metronomic oral doses of cyclophosphamide for the treatment of patients with surgically resected adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Has a history of surgically resected and pathologically proved AJCC stage I or stage II adenocarcinoma of the head, neck, or uncinate of the pancreas.
2. Cohorts 1, 3, 4 and 5: Have been a participant in Hopkins IRB protocol J0810, J1568, J15237 or J1766.
3. Cohort 2: Have never received any type of pancreatic cancer vaccine/immunotherapy, had the Whipple surgery within 18 months and completed the planned adjuvant chemotherapy and/or chemoradiation.
4. Cohorts 1, 3, 4 and 5: Received the last irradiated GM-CSF transfected allogeneic pancreatic cell lines Panc 10.05 and Panc 6.03 at least 6-12 months prior.
5. Has received the last anti-cancer therapy at least 28 days ago.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Has provided informed consent.
8. Has adequate hematologic function.(Hemoglobin ≥ 9 g/dL ANC ≥ 1500/mm3 Platelets ≥ 100,000 K/ mm3).
9. Has adequate renal function (Serum creatinine ≤ 2 mg/dL).
10. Has adequate hepatic function. (Bilirubin ≤ 2.0 mg/dl, unless known Gilbert's Syndrome; AST, ALT and amylase ≤ 2x upper limit of normal, Alk Phos ≤ 5x upper limit of normal).
11. Agree to use adequate birth control, if of childbearing potential.

Exclusion Criteria:

1. Has radiographic evidence of pancreatic cancer recurrence.
2. Has any documented history of autoimmune diseases including systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis, glomerulonephritis,or vasculitis.
3. Has any uncontrolled medical problems.
4. Has had systemic steroid therapy within 28 days before vaccine administration.
5. Has an anticipated need for systemic steroid therapy within 28 days after vaccine administration.
6. Has any evidence of active infections.
7. Is pregnant.
8. Has a history of another cancer (other than pancreatic cancer) or myeloproliferative disorders in the past five years except for treated non-melanoma skin cancer, superficial bladder cancer, or carcinoma in-situ of the cervix.
9. Has a history of noncompliance during previous vaccination cycles with study treatment and/or monitoring which is concerning for continued noncompliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-04-20 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2026-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laheru, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data entry and analysis is still ongoing.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (J0810 Arm A): Patients coming from J0810 (NCT00727441) Patients receive GVAX
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Cohort 1 (J0810 Arm B): Patients coming from J0810 (NCT00727441) Patients receive IV CY and GVAX
  Cyclophosphamide (CY): Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Cohort 1 (J0810 Arm C): Patients coming from J0810 (NCT00727441) Patients receive oral CY and GVAX
  Cyclophosphamide Pill: Cohort 1 patients (J0810 Arm C) will receive 50mg oral CY once a day starting 28 days prior to GVAX and for 28 days post-GVAX (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Cohort 3 (J1568): Patients coming from J1568 (NCT02451982) Patients receive IV CY and GVAX
  Cyclophosphamide: Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Cohort 4 (J15237): Patients coming from J15237 (NCT02648282) Patients receive IV CY and GVAX
  Cyclophosphamide: Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Cohort 5 (J1766): Patients coming from J1766 (NCT03153410) Patients receive IV CY and GVAX
  Cyclophosphamide: Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
Period: Overall Study
Arm/Group | Cohort 1 (J0810 Arm A) | Cohort 1 (J0810 Arm B) | Cohort 1 (J0810 Arm C) | Cohort 2 (Vaccine Naive) | Cohort 3 (J1568) | Cohort 4 (J15237) | Cohort 5 (J1766)
Started (Started = enrolled and received at least one dose of study drug) | 8 | 3 | 2 | 52 | 6 | 0 | 0
Completed (Completed = 10 years of treatment for Cohorts 1 and 2, and 5 years of treatment for Cohorts 3, 4, and 5) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 8 | 3 | 2 | 49 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled into Cohort 4 or Cohort 5
Groups:
- Cohort 1 (J0810 Arm B): Patients coming from J0810 (NCT00727441) Patients receive IV CY and GVAX
  Cyclophosphamide: Cohort 1 (J0810 Arm B), Cohort 3, Cohort 4, and Cohort 5 patients will receive 200mg/m^2 CY administered IV on day 0 of each Cycle (every 6 months). Cohort 2 patients will receive 200mg/m^2 CY administered IV on Day 0 of the first 3 cycles (every 28 days) and Day 0 of subsequent Cycles (every 6 months).
  GVAX Pancreas Vaccine: Cohort 1, 3, 4, and 5 patients will receive GVAX on day 1 of each Cycle (every 6 months). Cohort 2 patients will receive GVAX on Day 1 of the first 3 cycles (every 28 days) and Day 1 of subsequent Cycles (every 6 months).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (J0810 Arm A) | Cohort 1 (J0810 Arm B) | Cohort 1 (J0810 Arm C) | Cohort 2 (Vaccine Naive) | Cohort 3 (J1568) | Cohort 4 (J15237) | Cohort 5 (J1766) | Total
Number analyzed (Participants) | 8 | 3 | 2 | 52 | 6 | 0 | 0 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 0 | 35 | 2 | 0 | 0 | 45
  >=65 years | 3 | 0 | 2 | 17 | 4 | 0 | 0 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 24 | 4 | 0 | 0 | 34
  Male | 5 | 2 | 0 | 28 | 2 | 0 | 0 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 7 | 3 | 2 | 52 | 6 | 0 | 0 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Drug-Related Adverse Events (AEs) Requiring Treatment Discontinuation
Description: Safety as measured by local and systemic toxicity according to NCI CTCAE v 3.0
Time Frame: 121 Months
Population: No patients were enrolled into Cohort 4 or Cohort 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (J0810 Arm A) | Cohort 1 (J0810 Arm B) | Cohort 1 (J0810 Arm C) | Cohort 2 (Vaccine Naive) | Cohort 3 (J1568) | Cohort 4 (J15237) | Cohort 5 (J1766)
Number analyzed (Participants) | 8 | 3 | 2 | 52 | 6 | 0 | 0
Participants | 0 | 0 | 0 | 3 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Grade 3 or Above Drug-Related Adverse Events (AEs)
Description: Safety as measured by local and systemic toxicity according to NCI CTCAE v 3.0
Time Frame: 121 months
Population: No patients were enrolled into Cohort 4 or Cohort 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (J0810 Arm A) | Cohort 1 (J0810 Arm B) | Cohort 1 (J0810 Arm C) | Cohort 2 (Vaccine Naive) | Cohort 3 (J1568) | Cohort 4 (J15237) | Cohort 5 (J1766)
Number analyzed (Participants) | 8 | 3 | 2 | 52 | 6 | 0 | 0
Participants | 1 | 0 | 0 | 7 | 0 | 0 | 0

3. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS was measured as the time from date of surgery until pancreatic cancer recurrence or death. Disease status was monitored by radiologic scans done per standard of care. DFS was censored on the date of last radiologic scan for subjects without documentation of cancer recurrence or death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 131 months
Reporting Status: Not Posted, anticipated posting 2026-07

4. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the amount of time from date of surgery until death or end of follow-up. OS was censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 174 Months
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 121 months. All-cause mortality was evaluated for up to 133 months.
Description: No patients were enrolled into Cohort 4 or Cohort 5
Arm/Group | Cohort 1 (J0810 Arm A) | Cohort 1 (J0810 Arm B) | Cohort 1 (J0810 Arm C) | Cohort 2 (Vaccine Naive) | Cohort 3 (J1568) | Cohort 4 (J15237) | Cohort 5 (J1766)
All-Cause Mortality (participants affected / at risk) | 6/8 | 3/3 | 1/2 | 37/52 | 3/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/3 | 0/2 | 8/52 | 0/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/8 | 3/3 | 2/2 | 52/52 | 4/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (J0810 Arm A) (N=8) | Cohort 1 (J0810 Arm B) (N=3) | Cohort 1 (J0810 Arm C) (N=2) | Cohort 2 (Vaccine Naive) (N=52) | Cohort 3 (J1568) (N=6) | Cohort 4 (J15237) (N=0) | Cohort 5 (J1766) (N=0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholongitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FibroInflammatory lesion (pancreas) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subacute Peritoneal Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (J0810 Arm A) (N=8) | Cohort 1 (J0810 Arm B) (N=3) | Cohort 1 (J0810 Arm C) (N=2) | Cohort 2 (Vaccine Naive) (N=52) | Cohort 3 (J1568) (N=6) | Cohort 4 (J15237) (N=0) | Cohort 5 (J1766) (N=0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 7 (11) | 1 (1) | 0 (0) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 13 (27) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Edema Limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 37 (95) | 2 (4) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (4) | 0 (0) | 0 (0) | 12 (27) | 1 (1) | 0 (0) | 0 (0)
Flu-like Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (13) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 17 (26) | 1 (1) | 0 (0) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 26 (63) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 11 (18) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 24 (47) | 3 (6) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 2 (2) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 18 (53) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine Increase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Edema Face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema Tunk (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Pull (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT01088789/Prot_SAP_000.pdf